CLINICAL TRIAL: NCT03926832
Title: Prevalence of Obstructive Sleep Apnea Syndrome in Sarcoidosis and Impact of CPAP Treatment on Associated Fatigue Status
Acronym: SARCOIDOSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Pier Valerio Mari, Pulmonary and Critical Care Medicine (P/CCM) senior fellow, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2455
Record Dates: First submitted 2019-04-19; First posted 2019-04-25 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Sarcoidosis; Sleep Apnea, Obstructive; Fatigue
Keywords: CPAP
MeSH Terms: conditions — Sarcoidosis; Sleep Apnea, Obstructive; Fatigue | interventions — Continuous Positive Airway Pressure; Positive-Pressure Respiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Sarcoidosis (Experimental): Participants with Sarcoidosis. This arm will complete baseline questionnaires assessing daytime sleepiness (Epworth Sleepiness Scale - ESS) and fatigue (Fatigue Assessment Scale - FAS). All participants will perform home polygraphy and will be treated with CPAP for three months if moderate-to-severe OSA has been diagnosed and re-assessed with the same questionnaires along with a complete analysis of CPAP adherence by analyzing the compliance report of the device.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — Continuous positive airway pressure (CPAP) is the gold standard for Obstructive Sleep Apnea Syndrome (OSAS) management when moderate-to-severe. Subjects with OSA will be trained in the use of CPAP and will be instructed to use it every night for 3 months. These subjects will then return for a post-treatment completion of questionnaires (ESS and FAS) and compliance analysis.
  Other Names: positive airway pressure; positive pressure ventilation

SUMMARY:
Sarcoidosis is a multisystemic granulomatous disease that affects individuals worldwide without known pathogenesis, and the role of comorbidities has not been fully assessed in the scientific literature. An increased incidence of Obstructive Sleep Apnea Syndrome (OSAS) has been described in Sarcoidosis although this association has not been explained yet and no data is available about the effect of treatment with Continuous Positive Airway Pressure (CPAP) in Sarcoidosis. Also, patients affected by Sarcoidosis usually experience a state of physical and mental weariness called fatigue and reported in approximately 60-80% sarcoid patients and thought to be a consequence of inflammatory mediators but the high prevalence of OSAS could be a remarkable bias in clinical evaluation because fatigue is also strongly associated with sleep disorders.

Thus, there is a real need for assessing not only the real prevalence of OSAS in Sarcoidosis but also the effect of CPAP treatment on fatigue status experienced by sarcoidotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a definite diagnosis of sarcoidosis according to international ATS and WASOG guideline

Exclusion Criteria:

* Ongoing CPAP treatment
* Psychiatric disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-04-27 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Obstructive Sleep Apnea | Day 1
  Number of participants for whom polysomnography has shown an Apnea Hypopnea Index (AHI) more than 5 events/hour. Mild OSA is defined as AHI between 5 and 15 events/hour. Moderate OSA is defined as AHI between 15 and 30 events/hour. Severe OSA is defined as AHI more than 30 events/hour.

SECONDARY OUTCOMES:
Impact of Continuous Positive Airway Pressure (CPAP) treatment on fatigue associated status | Day 1, month 3 of CPAP treatment
  Change of "Fatigue Assessment Scale" (FAS) questionnaire result after the start of CPAP treatment in moderate-to-severe OSA patients affected by sarcoidosis. The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue. The minimal important difference is defined as a reduction of at least 4 points or 10% of baseline value.
Impact of Continuous Positive Airway Pressure (CPAP) treatment on daytime sleepiness | Day 1, month 3 of CPAP treatment
  Change of "Epworth Sleepiness Scale" (ESS) questionnaire result after the start of CPAP treatment in moderate-to-severe OSA patients affected by sarcoidosis. Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-1-2-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. A result more than 10 is suggestive of daytime sleepiness. The minimal important difference is defined as a reduction of at least 2 points of baseline value.
Compliance to CPAP treatment | 3 month post CPAP treatment
  Evaluate the treatment compliance of Sarcoidosis patients affected by moderate-to-severe OSA to CPAP therapy. Good CPAP compliance is defined as using the device for an average of more than 4 hours per night and at least 70% of total nights. Poor CPAP compliance is defined as using the device for an average of less than 4 hours per night and less than 70% of total nights. No compliance to CPAP treatment is defined if a patient refused to start CPAP treatment. Data about average time, percentages of device use during treatment will be determined analyzing the compliance report of the device based on integrated CPAP SD card data storage.
Baseline evaluation of fatigue status | Day 1
  Baseline assessment of fatigue status using the questionnaire "Fatigue Assessment Scale" (FAS). The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue.
Baseline evaluation sleepiness | Day 1
  Baseline assessment of sleepiness status using the questionnaire "Epworth Sleepiness Score" (ESS). The total score ranges from 0 to 24. Respondents are asked to rate, on a 4-point scale (0-1-2-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. A result in ESS score more than 10 is suggestive for daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Richeldi, MD, PhD, Study Director — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Policlinico Universitario Agostino Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No